CLINICAL TRIAL: NCT01285739
Title: Eight-year Follow up in Tracheostomized COPD Patients Undergoing Domiciliary Non Invasive Mechanical Ventilation.
Brief Title: Tracheostomized COPD Patients and Non Invasive Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Ercole Zanotti, MD, Fondazione Salvatore Maugeri
Other Study IDs: MS-12-2010
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2010-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Pulmonary Disease, Chronic Obstructive.; Tracheostomy.; Invasive Mechanical Ventilation.; Non-Invasive Mechanical Ventilation.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Leukocyte Count; Biomarkers; X-Rays; Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, tracheobronchial aspirate (TBA)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NIMV COPD: Patients with chronic obstructive pulmonary disease (COPD), who underwent tracheostomy for acute respiratory failure and who were discharged with tracheostomy but in domiciliary non invasive ventilation
  Interventions: Other: WBC, biomarkers, TBA, chest X ray
- IMV COPD: Patients with chronic obstructive pulmonary disease (COPD), who underwent tracheostomy for acute respiratory failure and who were discharged in domiciliary invasive mechanical ventilation (IMV)
  Interventions: Other: WBC, biomarkers, TBA, chest X ray

INTERVENTIONS:
Other: WBC, biomarkers, TBA, chest X ray — The above cited parameters were recorded and investigated every six months; chest X ray when needed.
  Other Names: PCT; CRP
  Groups: NIMV COPD
Other: WBC, biomarkers, TBA, chest X ray — The above cited parameters were recorded and investigated every six months; chest X ray when needed.
  Other Names: PCT; CPR
  Groups: IMV COPD

SUMMARY:
The purpose of this study was to determine occurrence of ventilator associated pneumonia (VAP) in tracheostomized patients with COPD discharged in invasive mechanical ventilation (IMV) compared to patients with CPOPD discharged with tracheostomy but in non invasive mechanical ventilation (NIMV).

DETAILED DESCRIPTION:
Acute respiratory failure due to COPD is often treated with invasive mechanical ventilation through endotracheal intubation, followed by placement of a endotracheal canula. However, invasive ventilation is at risk of infective complications and is difficult to manage at home. In particular, invasive mechanical ventilation may be associated with ventilator associated pneumonia (VAP). VAP is usually suspected when the individual develops a new or progressive infiltrate on chest radiograph, leukocytosis, and purulent tracheobronchial secretions. When possible, we tried to put these tracheotomized patients in non invasive mechanical ventilation (NIMV)to avoid VAP. This population was followed for eight consecutive years and compared with patients in invasive home mechanical ventilation (IMV).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* Tracheostomy
* Need of domiciliary invasive / non invasive ventilation

Exclusion Criteria:

* Patients with COPD weaned from invasive / non invasive mechanical ventilation
* Lack of tracheostomy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort was selected from patients admitted to Weaning Center. Patients weaned from invasive mechanical ventilation but who needed to keep endotracheal canula were enrolled for the study. Patients with COPD, tracheostomized and in domiciliary invasive mechanical ventilation was the control group.
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2002-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
ventilator associated pneumonia (VAP) | six months
  VAP is usually suspected when the individual develops a new or progressive infiltrate on chest radiograph, leukocytosis, and purulent tracheobronchial secretions. Therefore white cell blood (WBC)count, procalcitonine (PCT), C-reactive protein (CRP) and tracheobronchial aspirate (TBA) were collected every 6 months. Chest X ray was performed only when a clinical suspect of VAP was advanced.

SECONDARY OUTCOMES:
Blood gas analysis | Six months
  Blood gas analysis
Care givers involvement | Six months
  Through a dedicated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ercole Zanotti, MD, Principal Investigator — Fondazione Salvatore Maugeri
Locations (1):
- Weaning Center - Fondazione Salvatore Maugeri IRCCS, Montescano, Pavia, Italy